CLINICAL TRIAL: NCT01535911
Title: Pilot Study of a Metabolic Nutritional Therapy for the Management of Primary Brain Tumors
Acronym: Ketones
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Sparrow Health System (Other)
Responsible Party: Principal Investigator, Kenneth Schwartz, MD, Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-452FS
Record Dates: First submitted 2012-02-03; First posted 2012-02-20 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma
Keywords: ketogenic diet; brain tumors
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Obsrvational study adding ketogenic diet to standard initial treatment of glioblastom multiforme (Experimental): Add ketogenic diet to standard tx of glioblastoma multiforme. After patients have recovered from surgical intervention patients are given a ketogenic diet along with standard of care, radiation and temozolomide treatments. The ketogenic diet is modified by dietitians based on twice daily measurements of blood ketone levels.
  Interventions: Other: Energy restricted Ketogenic Diet (ERKD) (Metabolic Nutritional Therapy)

INTERVENTIONS:
Other: Energy restricted Ketogenic Diet (ERKD) (Metabolic Nutritional Therapy) — Adult subjects with newly diagnosed glioblastoma will be referred to the study. Residual tumor size will be determined using MRI imaging. Subjects will be placed on ERKD while they are being treated with radiation therapy and standard of care chemotherapy. After completion of radiation therapy, tumor size will be determined using MRI. If the tumor has decreased in size or remained the same (stable disease), the subjects will be continued on the ERKD for an additional 6 weeks. Total calories consumed by each subject will be targeted to 20 to 25 kcal/kg/day. If the tumor has decreased in size or the size has remained the same then subjects will be continued on the ERKD for as additional 6 weeks and a repeat MRI will be obtained.
  Other Names: Ketogenic diet

SUMMARY:
This study will look at the effects, good and/or bad, of treating primary brain cancers with diet therapy using an energy restricted ketogenic diet (ERKD) that uses food. An energy restricted ketogenic diet is a diet designed to keep blood sugars in the low range of normal while at the same time increasing the blood concentration of metabolic break down products called ketones. This diet is currently used to treat children with uncontrollable seizures. This diet is well tolerated by the children with minimal side effects reported after using the diet for years.

* The main purpose of this study is to find out whether or not the energy restricted ketogenic diet will help patients with primary brain cancer by either decreasing the size of the cancer or by keeping the cancer from growing.
* Another reason for doing this study is to learn about the side effects associated with the energy restricted ketogenic diet in patients with primary brain cancer.

DETAILED DESCRIPTION:
Summary: The current standard of care for glioblastoma multiforme (GBM), the most common primary brain tumor in adults, includes surgical resection, radiation and chemotherapy. Survival rarely exceeds 18 months. The investigators propose to test the hypothesis that brain tumor cells are unable to utilize ketones as a source of energy when deprived of glucose, due to mitochondrial dysfunction, whereas normal glia and neurons can survive this metabolic stress. A nutritionally adequate but energy restricted, ketogenic diet (ERKD) to deprive brain tumors of energy and resulting in death of glioma cells is promising. ERKD-based therapy to manage brain cancer is both biologically plausible and supported by data in animal models. A multidisciplinary team of oncologists, registered dietitians, and physiologists will implement an ERKD therapy in newly diagnosed GBM subjects. After initial maximal tumor excision, ERKD therapy will be initiated for subjects during a one week inpatient admission to Sparrow Hospital or as a local outpatient and supervised by registered dietitians experienced in implementing this therapy.The ERKD will continue as adjunctive therapy along with radiation therapy and standard of care chemotherapy. The supervised ERKD will continue for an additional 6 weeks after completion of radiation therapy along with the standard of care chemotherapy. The objective of this trial is to determine whether the ERKD decreases tumor size or results in no recurrence in individuals with GBM as measured by serial MRI imaging. Enzymes and signaling pathways that regulate metabolism and cell growth will be assessed in initial and post-ERKD tumors using standard biochemical approaches.

ELIGIBILITY:
* Inclusion Criteria:
* Adult subjects over age 18 with biopsy proven GBM diagnosis
* Measurable disease after standard therapies
* Eastern Cancer Oncology Group performance status < or =2; and
* Life expectancy >3 months.

Exclusion Criteria:

* Diagnosis of diabetes mellitus that is being treated by medication
* Concomitant use of glucocorticosteroids
* Cholecystectomy within 1 year prior to study entry
* Inability to adhere to or tolerate dietary protocol
* Active malignancy other than primary brain tumor requiring therapy
* Participation in an investigational study within 2 weeks prior to study entry; Major co-morbidities such as liver, kidney or heart failure that in the judgment of the investigators would disqualify the subject from the trial
* Pregnancy
* Inability to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
MRI imaging will be used to measure changes in brain tumor size. | 6 weeks after completion of radiation therapy
  Results of the metabolic therapy will be assessed by comparing MRI images obtained at the beginning of the study with those after completion of radiation therapy and after an additional 6 weeks of metabolic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Schwartz, MD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University/Sparrow Hospital, East Lansing, Michigan, United States

REFERENCES:
- [Background] Seyfried TN, Marsh J, Shelton LM, Huysentruyt LC, Mukherjee P. Is the restricted ketogenic diet a viable alternative to the standard of care for managing malignant brain cancer? Epilepsy Res. 2012 Jul;100(3):310-26. doi: 10.1016/j.eplepsyres.2011.06.017. Epub 2011 Aug 31. PMID 21885251
- [Derived] Schwartz K, Chang HT, Nikolai M, Pernicone J, Rhee S, Olson K, Kurniali PC, Hord NG, Noel M. Treatment of glioma patients with ketogenic diets: report of two cases treated with an IRB-approved energy-restricted ketogenic diet protocol and review of the literature. Cancer Metab. 2015 Mar 25;3:3. doi: 10.1186/s40170-015-0129-1. eCollection 2015. PMID 25806103